CLINICAL TRIAL: NCT05299502
Title: Promoting Healthy Eating in Early Pregnancy in Women at Risk of Gestational Diabetes Mellitus: Does it Improve Glucose Homeostasis?
Brief Title: Healthy Eating in Women at Risk of Gestational Diabetes
Acronym: SAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other)
Responsible Party: Principal Investigator, Anne-Sophie Morisset, Principal Investigator, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-6100
Record Dates: First submitted 2022-02-28; First posted 2022-03-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes; Pregnancy Complications
Keywords: Nutrition; Healthy Eating; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Intervention (Experimental): Intervention promoting healthy eating by a Registered Dietitian.
  Interventions: Behavioral: Nutritional Intervention
- Standard Care (No Intervention): Women will have their usual medical pregnancy follow-ups by their MDs without access to nutritional care.

INTERVENTIONS:
Behavioral: Nutritional Intervention — 4 individual 1-hour in person (or virtual, according to potential public health restrictions and patients' preference) motivational interviews (12, 18, 24 and 30 weeks) with a registered dietitian will be conducted to elaborate S.M.A.R.T. (Specific,Measurable, Attainable, Relevant, Timely) goals regarding diet, based on the 2019 Canada's Food Guide. Between those individual follow-ups, 4 phone calls with the registered dietitian will be provided (15, 21, 27, 33 weeks). Throughout the study, 10 informative nutritional video clips will also be provided. Participants receiving the intervention will have access to an online Facebook private community to discuss and share experiences, thus maintaining motivation and providing social support.
  Arms: Nutritional Intervention

SUMMARY:
Healthy eating during pregnancy has favorable effects on markers related to diabetes (glucose tolerance) and is associated with lower gestational diabetes mellitus (GDM) risk. The cornerstone of GDM treatment is nutrition therapy but the latter often starts late in pregnancy and thus may not have the expected effects on glucose tolerance. What if an intervention promoting healthy eating was initiated at the beginning of pregnancy in all women at risk, would it improve glucose homeostasis? To answer this important question, the investigators will perform a randomized controlled trial in 150 pregnant women. Women receiving the nutritional intervention will be compared to a control group receiving standard care. The nutritional intervention, which will start in the first trimester, is based on the 2019 Canada's Food Guide and is composed of 4 individual sessions with a registered dietitian (12, 18, 24 and 30 weeks). Between those follow-ups, informative nutritional web capsules and phone calls with the registered dietitian will be provided. To ensure that the women remain motivated and receive social support, a private Facebook group will be used. The investigators hypothesize that the nutritional intervention will be effective at improving glucose homeostasis. The investigators expect the results will show the importance of nutritional care starting early in pregnancy in women at risk of GDM.

DETAILED DESCRIPTION:
Individuals will participate in three on-site research visits during which a 2-hour oral glucose tolerance test will be performed. At each of these trimesters and 3 months after the delivery, participants will also complete three validated web-based 24-h recalls from which diet quality will be assessed. Subjects will be randomized to two arms after the first oral glucose tolerance test at the first visit. For all participants, on-site follow-ups by the research team will occur at each trimester and 1 virtual follow-up will be done 3 months after delivery for both groups. The total duration of participation for all is approximately 9 months.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 14 gestational weeks;
* Singleton pregnancy;
* At risk of GDM According to Diabetes Canada (being 35 years of age or older or from a high-risk group (African, Arab, Asian, Hispanic, Indigenous, or South Asian) or having a BMI ≥ 30 kg/m2, prediabetes, GDM in a previous pregnancy, given birth to a baby that weighed more than 4 kg, a parent, brother or sister with type 2 diabetes, polycystic ovary syndrome or acanthosis nigricans (darkened patches of skin).

Exclusion Criteria:

* Having a diabetes diagnosis in the 1st trimester;
* Pre-existing diabetes mellitus;
* Diseases requiring active nutritional treatment or influencing glucose metabolism (including previous bariatric surgery);
* Taking part in a nutritional intervention program;
* Corticosteroid use;
* Previous or current diagnosis of an eating disorder;
* Inability to give informed consent;
* Inability to communicate in French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | Changes from the 1st to the 3rd trimester
  Measured after a 12-hour fast.

SECONDARY OUTCOMES:
Post-prandial plasma glucose | Changes from the 1st to the 3rd trimester
  Measured 60 and 120 minutes during a 2-hour Oral Glucose Tolerance Test
Glycemic response | Changes from the 1st to the 3rd trimester
  Using incremental area under the curve for the blood glucose during a 2-hour Oral Glucose Tolerance Test
Hepatic insulin sensitivity | Changes from the 1st to the 3rd trimester
  Homeostasis Model Assessment of Insulin Sensibility
Hepatic and peripheral insulin sensitivity index | Changes from the 1st to the 3rd trimester
  Matsuda index
Beta-cell function index | Changes from the 1st to the 3rd trimester
  Disposition index: Matsuda index*insulinogenic index
Gestational Diabetes Mellitus diagnosis | End of pregnancy
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Morisset, RD, PhD, Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- CHU de Québec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier E, Plante AS, Lemieux P, Robitaille J, Lemieux S, Desroches S, Belanger-Gravel A, Maheux-Lacroix S, Weisnagel SJ, Demers S, Camirand Lemyre F, Boulet M, Baillargeon JP, Morisset AS. Promoting healthy eating in early pregnancy in individuals at risk of gestational diabetes mellitus: does it improve glucose homeostasis? A study protocol for a randomized control trial. Front Nutr. 2024 Jan 19;10:1336509. doi: 10.3389/fnut.2023.1336509. eCollection 2023. PMID 38312142